CLINICAL TRIAL: NCT04013269
Title: Effect of the CytoSorb Adsorber on Hemodynamic, Immunological and Pharmacokinetic Parameters in Refractory Septic Shock
Brief Title: Adjuvant Therapy With CytoSorb in Refractory Septic Shock
Acronym: ACYSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACYSS; DRKS00015483 (Registry Identifier: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2019-06-15; First posted 2019-07-09 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Septic Shock
Keywords: Sepsis; Critically ill; Intensive care medicine; CytoSorb; Hemoadsorption; Pharmacokinetic
MeSH Terms: conditions — Shock, Septic; Sepsis; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CytoSorb-Therapy (Active Comparator): Therapy of septic shock using guideline directed standard of care, including continuous renal replacement therapy in combination with haemadsorption using CytoSorb-Adsorber
  Interventions: Device: CytoSorb-Therapy
- Standard of care (No Intervention): Therapy of septic shock using guideline directed standard of care, including continuous renal replacement therapy

INTERVENTIONS:
Device: CytoSorb-Therapy — Additional use of Cytosorb-Adsorber in patients with septic shock and need for continuous renal replacement therapy
  Arms: CytoSorb-Therapy

SUMMARY:
This prospective randomized single center study investigates to what extent the removal of elevated cytokine levels by hemoadsorption has a positive effect on the treatment of patients in septic shock by stabilizing the circulatory situation.

DETAILED DESCRIPTION:
The term "sepsis" refers to a clinical syndrome in which a dysregulation of the host's inflammatory reaction to infection leads to a life-threatening of organ dysfunctions. Sepsis and septic shock are major causes of death in intensive care units worldwide.

The clinical picture of septic shock, the most severe form of sepsis, leads to uncontrolled production and release of a large number of proinflammatory cytokines and mediators, the "cytokine storm". Septic shock is accompanied by a massive increase in mortality of up to 60%.

This high mortality rate is due to a lack of current treatment options. The early recognition of the disease and its immediate treatment are decisive for successful therapy and the survival of those affected. The most important therapeutic steps, apart from focus control by antibiotics and surgical intervention, are the stabilization of the affected organ systems, in particular the circulatory system and the respiratory system. As an extracorporeal and non-specific procedure for the interruption of the cytokine storm, hemoadsorption by means of CytoSorb adsorbers may be an intervention, which has already demonstrated its basic effectiveness in the treatment of septic and cardiosurgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Refractory septic shock
* Need for Norepinephrine ≥ 0.25 µg/kg/min
* IL6 ≥ 1000 ng/l
* Indication for CRRT

Exclusion Criteria:

* Sepsis due to pulmonary or urogenital causes
* Onset of septic shock longer than 36 hours
* Liver cirrhosis Child Pugh C
* "do not resuscitate"-order
* expected survival < 14 days
* participation in another interventional trial
* Pregnancy or breastfeeding
* Lack of consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a reduction of catecholamine dose of at least 25% within the first 48 hours of treatment | 48 hours
  Percentage of patients with a reduction of catecholamine dose of at least 25% compared to baseline for at least 6 hours within the first 48 hours of treatment.

SECONDARY OUTCOMES:
Change in organ dysfunction | 10 days
  Change in organ dysfunction based on "Sequential Organ Failure Assessment" (SOFA) Score The SOFA score is made of 6 variables, each representing an organ system. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure) The worst physiological variables were collected serially every 24 hours of a patient's ICU admission. The "worst" measurement was defined as the measure that correlated to the highest number of points. The SOFA score ranges from 0 to 24.
Lactate clearance | 10 days
  Improving lactate clearance by lowering serum lactate levels
Renal replacement therapy | 10 days
  Time with need for renal replacement therapy
Percentage of patients with a reduction of catecholamine dose of at least 25% within the first 24 hours of treatment | 24 hours
  Percentage of patients with a reduction of catecholamine dose of at least 25% compared to baseline for at least 6 hours within the first 48 hours of treatment.
End of septic shock | 10 days
  Time until shock resolution
ICU length of stay | 90 days
  ICU length of stay
Time on mechanical ventilation | 10 days
  Time on mechanical ventilation
Cumulative catecholamine dose | 10 days
  Cumulative catecholamine dose
Overall and ICU mortality | 90 days
  Overall and ICU mortality
Serum levels of administered anti-infectives | 3 days
  Serum drug Levels of pre and post filter and adsorber system on day 1-3 while CytoSorb therapy (sampling: t 0, 1, 2, 6, 8, 12, 24 h after CytoSorb initiation)
Change of plasma Interleukin-6 (IL6) level | 10 days
  Change of plasma Interleukin-6 (IL6) level
Change of plasma Interleukin-10 (IL10) level | 10 days
  Change of plasma Interleukin-10 (IL10) level
Change of plasma Procalcitonin (PCT) level | 10 days
  Change of plasma Procalcitonin (PCT) level
Change of HLA-DR level | 10 days
  Change of HLA-DR (Human Leukocyte Antigen - DR isotype) level of monocytes
Change of TNF alpha level after ex-vivo stimulation | 10 days
  Change of TNF-alfa level (Tumor Necrosis Factor alpha) level after LPS (Lipopolysaccharides) stimulation as sign of monocytic immunocompetence

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, MD, Principal Investigator — University Hospital Hamburg-Eppendorf, Department of Intensive Care Medicine
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taeb AM, Hooper MH, Marik PE. Sepsis: Current Definition, Pathophysiology, Diagnosis, and Management. Nutr Clin Pract. 2017 Jun;32(3):296-308. doi: 10.1177/0884533617695243. Epub 2017 Mar 17. PMID 28537517
- [Background] Friesecke S, Stecher SS, Gross S, Felix SB, Nierhaus A. Extracorporeal cytokine elimination as rescue therapy in refractory septic shock: a prospective single-center study. J Artif Organs. 2017 Sep;20(3):252-259. doi: 10.1007/s10047-017-0967-4. Epub 2017 Jun 6. PMID 28589286
- [Background] Garau I, Marz A, Sehner S, Reuter DA, Reichenspurner H, Zollner C, Kubitz JC. Hemadsorption during cardiopulmonary bypass reduces interleukin 8 and tumor necrosis factor alpha serum levels in cardiac surgery: a randomized controlled trial. Minerva Anestesiol. 2019 Jul;85(7):715-723. doi: 10.23736/S0375-9393.18.12898-7. Epub 2018 Nov 22. PMID 30481999
- [Background] Kogelmann K, Jarczak D, Scheller M, Druner M. Hemoadsorption by CytoSorb in septic patients: a case series. Crit Care. 2017 Mar 27;21(1):74. doi: 10.1186/s13054-017-1662-9. PMID 28343448
- [Background] Bayer O, Reinhart K, Kohl M, Kabisch B, Marshall J, Sakr Y, Bauer M, Hartog C, Schwarzkopf D, Riedemann N. Effects of fluid resuscitation with synthetic colloids or crystalloids alone on shock reversal, fluid balance, and patient outcomes in patients with severe sepsis: a prospective sequential analysis. Crit Care Med. 2012 Sep;40(9):2543-51. doi: 10.1097/CCM.0b013e318258fee7. PMID 22903091